CLINICAL TRIAL: NCT05882552
Title: The Accuracy of Applying the Tilted Gaze Target Test in the Examination of Children With Superior Oblique Muscle Palsy
Brief Title: Tilted Gaze Target Test in the Examination of Children With Superior Oblique Muscle Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2023018
Record Dates: First submitted 2023-05-06; First posted 2023-05-31 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Children With Torticollis
Keywords: tilted gaze; superior oblique muscle palsy; strabismus; diagnosis; projection
MeSH Terms: conditions — Strabismus; Disease

STUDY DESIGN:
Intervention Model Description: The enrolled study participants will be randomly assigned to two groups and undergo a crossover design in which they will sequentially undergo the tilted gaze target test and conventional examination methods, including oculomotor examination, Bielschowsky tilt test, alternate prism cover test, prism adaptation test, and monocular cover test.
Who Masked: Participant, Care Provider, Investigator
Masking Description: During the procedure, the participants will not be informed of the results of the gaze tilt test. The tilted gaze target test will be conducted by a professional ophthalmologist who is not involved in the consultation and is unaware of the actual diagnosis of the study participants. The investigators will ensure that the normal consultation process is followed without being informed of the results of the gaze tilt test. The statistical analysis will be performed by a third-party outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tilted Gaze Target Test+Conventional Examinations (Experimental): Tilted gaze target test is before conventional examination
  Interventions: Diagnostic Test: Tilted Gaze Target Tast; Diagnostic Test: Conventional Examination Methods
- Conventional Examinations +Tilted Gaze Target Test (Active Comparator): Conventional examination is before tilted gaze target test
  Interventions: Diagnostic Test: Tilted Gaze Target Tast; Diagnostic Test: Conventional Examination Methods

INTERVENTIONS:
Diagnostic Test: Tilted Gaze Target Tast — Tilted gaze target tast is playing a small animated video with a visual mobile device at a distance of 33 cm and 3 m, respectively, to determine the optimal angle of head position improvement and the spatial tilt angle of the screen relative to the orthostatic position.It will be conducted during the first visit. Preoperative intervention will also be conducted before surgery. Postoperative interventions will be conducted at one day, one month, and six months after surgery.
Diagnostic Test: Conventional Examination Methods — The conventional examination methods include oculomotor examination, Bielschowsky head tilt test, alternate prism cover test, prism adaptation test, and monocular cover test. They will be conducted during the first visit. Preoperative intervention will also be conducted before surgery.Postoperative interventions will be conducted at one day, one month, and six months after surgery.

SUMMARY:
This study is a prospective, randomized, double-blind cohort study aimed at assessing the accuracy of the preoperative tilted gaze target test in predicting the degree of improvement in compensatory head position after surgery in children with superior oblique muscle palsy.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind cohort study conducted from May 2023 to April 2024. The study aims to evaluate the effectiveness of a non-human contact gaze tilt test in the diagnosis of children with superior oblique Muscle Palsy. Patients who met the inclusion criteria for outpatient and inpatient ophthalmic surgery for strabismus and pediatric ophthalmology were enrolled after signing a written informed consent. The gaze tilt test was added to the normal treatment process and performed by a professional ophthalmologist who was not involved in the treatment process. The test involved playing a small animated video with a visual mobile device at a distance of 33 cm and 3 m, respectively, to determine the optimal angle of head position improvement and the spatial tilt angle of the screen relative to the orthostatic position. A third-party analysis of the data was performed to identify myotonic and oculocutaneous tilts and compared with the results of the conventional test. The study aims to clarify the authenticity, reliability, and practicality of the gaze object tilt test in diagnosing and treating oculocutaneous squint.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 and 8 years old.
* History of torticollis less than 5 years.
* Ability to cooperate with basic examinations at the Tianjin Ophthalmology Strabismus and Pediatric Ophthalmology Clinic.
* Complete clinical information available.
* Signed informed consent.

Exclusion Criteria:

* Both eyes cannot look at the same time or alternately
* Children with ocular disease other than oculomotor eye disease.
* Clearly defined systemic developmental abnormalities: Down syndrome, microcephaly, autism, Leber syndrome, central visual impairment, etc.
* Children who cannot cooperate with the examination due to age or other reasons.

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The accuracy of test in predicting the degree of improvement in head position after surgery | 6 Months
  Pearson correlation and paired sample difference analyses were conducted to compare the results of the preoperative gaze object tilt test (tilted post-tilt head angle/untilted head angle) with the postoperative head angle measurements taken at 1 day, 1 month, and 6 months, relative to the preoperative untilted head angle.

SECONDARY OUTCOMES:
Comparison with the traditional combined diagnosis of monocular masking, eye movement and Bielschowsky head-tilting test，the positive predictive value of tilt test in the diagnosis and treatment of oculomotor-derived torticollis | 1Week
  Positive predictive value= (True Positives / (True Positives + False Positives)) * 100
Comparison with the traditional combined diagnosis of monocular masking, eye movement and Bielschowsky head-tilting test，the negative predictive value of tilt test in the diagnosis and treatment of oculomotor-derived torticollis | 1Week
  Negative predictive value =(True Negatives / (True Negatives + False Negatives)) * 100

OTHER OUTCOMES:
The correlation between tilted gaze target test and Bielschowsky's head tilt test | 6 Months
  Pearson correlation and paired sample difference analyses were conducted to tilted gaze target test and Bielschowsky's head tilt test results
The correlation between the tilt angle and the degree of vertical and rotational strabismus | 6 Months
  Pearson correlation and paired sample difference analyses were conducted to the correlation between the tilt angle and the degree of vertical and rotational strabismus

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, Ph.D, Study Chair — Tianjin Eye Hospital; Xiaotong Li, M.D., Study Director — Tianjin Eye Hospital; Tiange Liu, MA.Sc, Principal Investigator — Nankai University; Zhen Li, MA.Sc, Principal Investigator — Nankai University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McLean JM. Direct Surgery of Underacting Oblique Muscles. Trans Am Ophthalmol Soc. 1948;46:633-51. No abstract available. PMID 16693495
- [Background] PARKS MM. Isolated cyclovertical muscle palsy. AMA Arch Ophthalmol. 1958 Dec;60(6):1027-35. doi: 10.1001/archopht.1958.00940081047008. No abstract available. PMID 13593934
- [Background] Hertle RW. Diagnosis of isolated cyclovertical muscle overaction using a modification of the Parks' Three-Step Test. Strabismus. 1993;1(3):107-20. doi: 10.3109/09273979309057131. PMID 21314550
- [Background] Khorrami-Nejad M, Akbari MR, Kangari H, Akbarzadeh Baghban A, Masoomian B, Ranjbar-Pazooki M. Abnormal Head Posture in Unilateral Superior Oblique Palsy. J Binocul Vis Ocul Motil. 2021 Jan-Mar;71(1):16-23. doi: 10.1080/2576117X.2020.1845561. Epub 2020 Dec 16. PMID 33326345
- [Background] Chung SA, Yim SY, Park A. Sternocleidomastoid muscle asymmetry in unilateral congenital superior oblique palsy. Eye (Lond). 2021 Jul;35(7):1954-1960. doi: 10.1038/s41433-020-01205-2. Epub 2020 Sep 30. PMID 32999476